CLINICAL TRIAL: NCT04752839
Title: Evaluation of the Psychosocial Impact on Health Professionals Exposed During the COVID 19 Coronavirus Pandemic
Brief Title: Evaluation of the Psychosocial Impact on Health Professionals Exposed During COVID 19 Coronavirus Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-40
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Psychological Stress; Psychosocial Impairment; Anxiety; Depression; Post Traumatic Stress Disorder; Coronavirus Infection; COVID
Keywords: Covid 19; Healthcare workers; Mental health
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Coronavirus Infections; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposed Workers: Workers who have been exposed during COVID 19 pandemic.

SUMMARY:
Application of a survey in electronic support to hospital professionals. This survey will include different demographics as well as questions from own elaboration about the different aspects related to the development of work during the health emergency. A third part will be included different validated scales for screening / diagnosis of different problems that can present those who are working in the Current situation. The different scales are the PHQ-9, GAD 7, ISI, and EIE-R. These scales address the different problems that have been seen that can introduce professionals, Depression, Anxiety, Insomnia and adaptation to stressors.

ELIGIBILITY:
Inclusion Criteria:

* Workers during COVID 19 pandemic at Hospital de la Creu i Sant Pau

Exclusion Criteria:

* No Exclusion Criteria, only the negative to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is made up of workers from the Hospital de la Santa Creu i Sant Pau.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder (GAD7) score. | Through study completion, an average of 1 year.
  This instrument has been created to serve as a screening in anxiety disorder widespread. It is composed of 7 Likert-type response items from 0 to 3 that include the symptoms and the disability associated with the disorder.7 For its correction, a total score is obtained from the sum of scores of all the items, which can range from 0 to 21.
  There are no established cut-off points for the Spanish version. In the original version, the authors propose a cut-off point of greater than or equal to 10. The version validated for the Spanish population will be used.
Insomnia severity Index (ISI) | Through study completion, an average of 1 year.
  The investigators will use the adaptation of Fernández Mendoza et al. It is made up of 7 items that evaluate the nature, severity and impact of insomnia. It is answered with a Likert-type scale that goes from 0 to 4, taking into account the last month.
  For its correction, a total score is obtained that ranges between 0 and 28. The proposed cut-off points of the original version are:
  * 0-7: no insomnia
  * 8-14: insomnia below the threshold
  * 15-21: clinical insomnia of moderate severity
  * 22-28: severe clinical insomnia
Patient Health Questionaire (PHQ-9) | Through study completion, an average of 1 year.
  This instrument is intended to aid the diagnosis of depression through the DSM-IV criteria, and to determine the severity of said disorder. It can also be used to observe the changes experienced by patients over time.
  It is made up of 9 items with Likert-type responses with values between 0 and 3 that refer to the last two weeks.
  For its correction, a total score is obtained that ranges between 0 and 27. The proposed cut-off points are:
  * 1-4: minimal depression
  * 5-9: mild depression
  * 10-14: moderate depression
  * 15-19: moderately severe depression
  * 20-27: severe depression The version validated for the Spanish population will be used
Perceived Stress Scale | Through study completion, an average of 1 year.
  The Perceived Stress Scale provides an overall measure of perceived stress in the last month evaluating the degree to which life situations are valued as stressful by people. 12 Specifically: the degree of subjective control over unpredictable or unexpected situations and the discomfort that accompanies the perceived lack of control. Originally it consists of 14 items (some of which are formulated in negative).
  Two dimensions have been considered (control and loss of control) although more restrictive criteria would require considering the one-dimensionality of the scale.
  The validated Spanish version will be used.
Impact of Event Scale Revised (IES-R) | Through study completion, an average of 1 year.
  This scale is conceptually based on Horowitz's two-factor theory and assesses the subjective discomfort that accompanies traumatic experiences. It is a self-administered scale, and consists of 22 items in the revised version. 7 items value intrusion 8 avoidance and 7 hyperactivation. The investigators will evaluate the post-traumatic stress symptomatology, and for that, the revised version in Spanish will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nickell LA, Crighton EJ, Tracy CS, Al-Enazy H, Bolaji Y, Hanjrah S, Hussain A, Makhlouf S, Upshur RE. Psychosocial effects of SARS on hospital staff: survey of a large tertiary care institution. CMAJ. 2004 Mar 2;170(5):793-8. doi: 10.1503/cmaj.1031077. PMID 14993174
- [Background] Maunder R, Hunter J, Vincent L, Bennett J, Peladeau N, Leszcz M, Sadavoy J, Verhaeghe LM, Steinberg R, Mazzulli T. The immediate psychological and occupational impact of the 2003 SARS outbreak in a teaching hospital. CMAJ. 2003 May 13;168(10):1245-51. PMID 12743065
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Fernandez-Mendoza J, Rodriguez-Munoz A, Vela-Bueno A, Olavarrieta-Bernardino S, Calhoun SL, Bixler EO, Vgontzas AN. The Spanish version of the Insomnia Severity Index: a confirmatory factor analysis. Sleep Med. 2012 Feb;13(2):207-10. doi: 10.1016/j.sleep.2011.06.019. Epub 2011 Dec 14. PMID 22172961
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Báguena M, Villarroya E, Beleña Á, Díaz A, Roldán C, Reig R. Propiedades Psycometricas de la Version Española de la Escala Revisionada de Impacto del Estresor (EIE-R). Anal y Modif Conduct. 2001;27(1997):581-604.